CLINICAL TRIAL: NCT02659579
Title: Evaluating the Effectiveness of the Reader Organisation's Get Into Reading Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Caroline Rowland (Other)
Responsible Party: Sponsor-Investigator, Caroline Rowland, Prof, University of Liverpool
Organization: University of Liverpool (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ES/M003752/1
Record Dates: First submitted 2016-01-07; First posted 2016-01-20 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Language Development
Keywords: Shared Book Reading; Vocabulary; Language Development; Young Children; Randomised Control Trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- The Reader Organisation's Shared Reading Programme (Experimental): In the Reader Organisation's Shared Reading Programme, parents and children will attend The Reader Organisation's weekly shared reading programme for 8 weeks. The programme consists of two different modules. Parents will attend 'Magical Storytimes' with their children, in which a collection of shared book reading sessions are led by a project worker. Parents will also attend sessions on their own ('Stories for you and Yours') in which they will be informed how to choose books and read interactively with their child.
  Interventions: Behavioral: The Reader Organisation's Shared Reading Programme
- Shared Reading control (Active Comparator): In the Shared Reading control parents and children will attend a weekly shared reading group at a library for 8 weeks where parents/children will read in a shared reading group which will be coordinated by a group facilitator.
  Interventions: Behavioral: Shared Reading control

INTERVENTIONS:
Behavioral: The Reader Organisation's Shared Reading Programme — In The Reader Organisation's Shared Reading Programme, parents and children will attend weekly shared book reading sessions for 8 weeks which focus predominately on how to read interactively with children.
  Arms: The Reader Organisation's Shared Reading Programme
Behavioral: Shared Reading control — Parents and children will attend a weekly shared reading group at a library for 8 weeks
  Arms: Shared Reading control

SUMMARY:
The investigators will evaluate the effectiveness of a parent-child shared reading intervention run by The Reader Organisation. The investigators will be asking parents and children across Liverpool to either (i) attend a weekly shared reading programme or (b) to attend a weekly children's reading group at a library. The investigators will look at how the reading groups affect children's language development, by comparing children's language development before having gone to these groups and after they have attended these groups.

DETAILED DESCRIPTION:
This is a Randomised Control Trial to test whether The Reader Organisation's Shared Reading Programme is more effective at improving the language development of children than a free library reading group. Intervention group: Fifty parents of children (3 to 4-years of age) will be recruited to take part in a 8 weeks long shared reading programme. The shared reading programme is comprised of two different modules: a) 'Magical Storytimes', in which a collection of shared book reading sessions are led by a project worker and b) 'Stories for You and Yours', in which parents will be taught how to choose books and read interactively with their child. Control group: Fifty further families, matched for age and background will be recruited to a reading control group and asked to attend a weekly shared reading group at a library where parents/children will read in a shared pre-school library reading group, coordinated by a group facilitator. Location: The Shared Reading Programme will take place in the child's nursery (in nurseries across Liverpool). Control group parents and children will attend a weekly reading group at a library. All standardised tests, for all children, will take place in the child's nursery. Language gains from pre- to post- intervention will be measured.

ELIGIBILITY:
Inclusion Criteria:

All families will be included unless they fit the exclusion criteria below.

Exclusion Criteria:

This is a study of typically developing English-learning children. The following exclusion criteria are designed to exclude families in which the target child is at risk of atypical or delayed language acquisition:

* Children born before 37 weeks gestation (premature)
* Children who weighed less than 5lb 9oz at birth (low birth weight)
* Children who have had an ear infection/glue ear for longer than 3 months, 4-6 ear infections within a 6 month period or another identified hearing problem (e.g. at newborn hearing screening)
* Children with an identified developmental disability (e.g. Cerebral Palsy, Autism Spectrum Disorder, Fragile X syndrome, Muscular dystrophy, Di George syndrome, Down's syndrome, Williams syndrome)
* Children with a hearing or visual impairment
* Children who hear another language (not English) for 1 day or more in a typical week (please note that this also excludes children of parents who do not speak English)
* Children whose parents have a learning disability which puts their children at risk of language delay and excludes the parents from giving informed consent on their own and on their children's behalf.

Ages: 36 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in baseline language skills: British Picture Vocabulary Scale: Third edition | Baseline and 4 weeks after intervention and 6 months after the intervention
  The British Picture Vocabulary Scale: Third edition (BPVS3) will be administered to children baseline, 4 weeks, and 6 months after intervention. The BPVS3 assesses a child's receptive vocabulary; for each question, the researcher says a word and the child responds by selecting a picture from four options that best illustrates the word's meaning.

SECONDARY OUTCOMES:
Change in baseline language skills: Clinical Evaluation of Language Fundamentals - Preschool 2 UK. | Baseline, 4 weeks after intervention and 6 months after the intervention
  The Clinical Evaluation of Language Fundamentals - Preschool 2 UK (CELF Preschool-2) will be administered to children at baseline, 4 weeks, and 6 weeks after intervention.The CELF Preschool-2 is a published measure of linguistic knowledge of individual children which measures a broad range of language skills in young children. Specifically, we will use three subset tests from the CELF Preschool-2. The "sentence structure" subset will measure the children's understanding of simple and complex sentence structures. A sentence is read to the child and the child chooses, from a set of pictures, which picture ''goes with'' that sentence.The "word structure" subset measures the children's understanding of simple and complex word structures. A sentence is read about a particular picture and the child is asked to finish the sentence.The "expressive vocabulary" subset evaluate a child's ability to label pictures of people, objects, and actions.
Parent Child Questionnaire | Baseline and 4 weeks after intervention
  The Parent Child Questionnaire contains 78 items and assesses: satisfaction with parenting, parent's interaction with and knowledge of his or her child, parent's perception of how he/she communicates with a child, parents' experience of disciplining their child, parent's ability to promote a child's independence and parents' attitudes about gender roles in parenting.
Family Questionnaire | Baseline
  The Family Questionnaire records relevant demographic information (e.g. socio-economic status, parents' education, family language use, ethnicity, children's medical history) that was devised for the Economic Social Research Council funded United Kingdom Communicative Development Inventory study. This allows us to create a composite individual socio-economic background variable using maternal education and household income in order to identify high and low socio-economic status families and to confirm that the participant children are typically developing monolinguals.
Family Reading Questionnaire | Baseline and 4 weeks after intervention
  The Family Reading Questionnaire examines frequency of storybook reading, reading requests and child library visits, number of books and children's books in the home, parental reading habits, reading onset, and frequency of parent teaching behaviours about reading, such as teaching about print knowledge (e.g. how often do you teach your child how to print words/read words?) questions about book choice (e.g. books read in the last week, child's favourite book).
Children's Title Checklist | Baseline and 4 weeks after intervention
  The Children's Title Checklist indirectly measure a child's storybook exposure by assessing the parent's knowledge of children's book titles (Children's Title Checklist). The Children's Title Checklist consists of 40 titles of popular children's books and 20 foils.
Children's Author Checklist | Baseline and 4 weeks after intervention
  The Children's Author Checklist indirectly measures a child's storybook exposure by assessing the parent's knowledge of authors. The Children's Author Checklist consists of 40 names of authors of popular children's books and 20 foils.
The Reader Organisation's Baseline Questionnaire | Baseline
  The Reader Organisation's Baseline Questionnaire assess parents' attitudes towards reading and barriers towards reading.
The Reader Organisation's Follow Up Questionnaire | 4 weeks after intervention
  The Reader Organisation's Follow Up Questionnaire assess parents' attitudes towards reading and barriers towards reading. Parents are also asked questions about their own experience of the intervention itself.
Leuven Scale during Dyadic Videoed Book-Reading Sessions | Baseline and 4 weeks after intervention
  The Leuven scale will be used to assess the child's active engagement during videoed dyadic book-reading sessions. There are 5 levels of engagements: extremely low (e.g. the child shows hardly any activity), low (e.g. the child shows some degree of activity which is often interrupted), moderate (e.g. the child is busy the whole time, but without real concentration), high (e.g. there are clear signs of involvement, but these are not always present to their full extent) and extremely high (e.g. during the observation of learning the child is continually engaged in the activity and completely absorbed in it).

CONTACTS AND LOCATIONS:
Overall Officials: Caroline F Rowland, PhD, Principal Investigator — University of Liverpool
Locations (1):
- Livepool Language Lab at the University of Liverpool, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
With the consent of participating adults, the data will be donated to the UK data archive.